CLINICAL TRIAL: NCT00024427
Title: An Open Label, Randomized, Controlled, Phase III, Multi-center, Clinical Trial Of PN401 With High Dose 5-Fluorouracil (5FU) Versus Gemcitabine For Treatment Of Patients With Advanced Pancreatic Cancer
Brief Title: Triacetyluridine and Fluorouracil Compared With Gemcitabine in Treating Patients With Unresectable Locally Advanced, or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wellstat Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068931; WELLSTAT-401.00.001; PRONEURON-401.00.001; UAB-0105; UAB-F010524008
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2010-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Pancreatic Cancer
Keywords: drug/agent toxicity by tissue/organ; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; uridine triacetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluorouracil — High dose 5-FU
  Other Names: 5-FU
Drug: gemcitabine hydrochloride — Normal dose to treat pancreatic cancer
  Other Names: Gemzar
Drug: triacetyluridine — 6 grams (12 tablets)
  Other Names: 2',3',5'tri-O-acetyluridine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different combinations may kill more tumor cells. Chemoprotective drugs such as triacetyluridine may protect normal cells from the side effects of chemotherapy. It is not yet known which chemotherapy regimen is more effective in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil plus triacetyluridine with that of gemcitabine in treating patients who have locally advanced or metastatic pancreatic cancer that cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with unresectable locally advanced or metastatic pancreatic cancer treated with triacetyluridine and high-dose fluorouracil vs gemcitabine.
* Compare the time to tumor progression, overall response rate, and response duration in patients treated with these regimens.
* Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to disease stage (II or III vs IV). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive high-dose fluorouracil (5-FU) IV over 30 minutes once weekly on weeks 1-3 followed by 1 week of rest. After each dose of 5-FU, patients receive oral triacetyluridine every 8 hours for a total of 8 doses. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 30 minutes once weekly on weeks 1-7 followed by 1 week of rest (course 1). Subsequent courses are given on weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 260 patients (130 per treatment arm) will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Unresectable locally advanced or metastatic disease

    * Stage II, III, or IV
* Measurable or evaluable disease
* No elevated tumor marker (CA 19-9) only
* No clinically significant third-space fluid accumulation (e.g., ascites or pleural effusion)
* No carcinoid, islet cell, or lymphoma of the pancreas
* No prior or concurrent brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.5 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT or AST less than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* No uncontrolled hepatic dysfunction

Renal:

* Creatinine less than 2.0 mg/dL
* No uncontrolled renal dysfunction

Cardiovascular:

* No uncontrolled cardiovascular disease requiring therapy, including the following:

  * Angina
  * Arrhythmias
  * Uncompensated cardiac failure
  * Myocardial infarction within the past 6 months

Pulmonary:

* No uncontrolled pulmonary dysfunction

Gastrointestinal:

* Able to take and/or retain oral medication
* No uncontrolled malabsorption syndrome or any other condition that would interfere with intestinal absorption

Other:

* No known allergy to fluorouracil (5-FU), gemcitabine, triacetyluridine, or any of their components
* No dihydropyrimidine-dehydrogenase deficiency
* No active uncontrolled infection
* No uncontrolled neurologic or psychiatric dysfunction
* No other malignancy except previously resected basal cell cancer or curatively resected stage I or less cervical cancer that has been disease free for at least 5 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy (including immunotherapy) for cancer

Chemotherapy:

* No prior chemotherapy for cancer other than as a radiosensitizer
* No prior 5-FU or gemcitabine other than as a radiosensitizer
* No prior triacetyluridine
* No other concurrent chemotherapy (including leucovorin calcium) for cancer

Endocrine therapy:

* No concurrent hormonal therapy for cancer
* Concurrent megestrol, oral contraceptives, or postmenopausal estrogen replacement therapy allowed

Radiotherapy:

* Prior radiotherapy allowed
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior resection of pancreas allowed

Other:

* At least 30 days since prior investigational drug or therapeutic device
* No other concurrent anticancer therapy
* No other concurrent investigational drugs or devices
* No concurrent drugs that would interact adversely with 5-FU or gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2001-02; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Open Label Randomized Phase 3 Multi-Center Trial of PN401 plus high dose 5-FU versus Gemcitabine in Advanced Pancreatic Cancer Patients | Disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Lenny Smith, MS, Study Chair — Wellstat Therapeutics
Locations (29):
- United States (26):
  - Brookwood Medical Center, Birmingham, Alabama
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - Northwest Oncology and Hematology Associates, Coral Springs, Florida
  - Florida Cancer Specialists - World Plaza, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Florida Oncology Associates - South Side, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Institute - New Port Richey, New Port Richey, Florida
  - St. Joseph's Hospital, Savannah, Georgia
  - Cancer Care Center, New Albany, Indiana
  - Cancer Center at Greater Baltimore Medical Center, Baltimore, Maryland
  - Wellstat Therapeutics, Gaithersburg, Maryland
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Queens Medical Associates, PC, Fresh Meadows, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Summit Oncology Associates, Akron, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase - Temple Cancer Center, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - Corpus Christi Cancer Center, Corpus Christi, Texas
- Canada (3):
  - Ottawa Regional Cancer Centre at Ottawa Hospital - General Campus, Ottawa, Ontario
  - Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec